CLINICAL TRIAL: NCT01585896
Title: Self-Help Group for the Treatment of Hoarding Disorder
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Kiara Timpano, Associate Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20111146
Record Dates: First submitted 2012-04-23; First posted 2012-04-26 (Estimated); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Hoarding Disorder
Keywords: Hoarding; Compulsive Hoarding; Self-Help
MeSH Terms: conditions — Hoarding Disorder; Hoarding | interventions — Self-Help Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Self-help group (Experimental): The facilitated self-help group, which represents an empirically supported intervention for hoarding (Frost et al., 2011).
  Interventions: Other: Self-Help Group

INTERVENTIONS:
Other: Self-Help Group — The facilitated self-help group may last approximately 13 sessions. This treatment represents an empirically supported intervention for hoarding (Frost et al., 2011), based on a Facilitator's Manual (Maxner et al., 2010), which is a treatment manual based on the book Buried in Treasures: Help for Compulsive Acquiring, Saving, and Hoarding (Tolin, Frost, & Steketee, 2007).

SUMMARY:
The proposed study aims to investigate the efficacy of a facilitated self-help group for the treatment of hoarding disorder. Eligible participants will take part in a facilitated self-help group. The investigators aim to investigate the effects of a self-help group on hoarding symptoms. The investigators hypothesize that participants will demonstrate decreased hoarding symptoms over time.

ELIGIBILITY:
Inclusion Criteria:

* clinically relevant symptoms of hoarding disorder

Exclusion Criteria:

* under 18
* psychotic disorders, bipolar disorder, substance abuse or dependence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-04 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Hoarding Rating Scale | 13 weeks
  Interviewer-rated measure of hoarding severity will be administered at Screening, Pre-Treatment, Mid-Treatment (approximately Week 7), Post-Treatment (approximately week 13), 1-month Follow-up The Hoarding Rating scale has a total score ranging from 0-40 with the higher score indicating higher symptoms of hoarding.

CONTACTS AND LOCATIONS:
Overall Officials: Kiara R Timpano, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of Miami Program for Anxiety, Stress, and OCD Research Webpage — https://paso.psy.miami.edu/research/index.html